CLINICAL TRIAL: NCT01297010
Title: Dexamethasone Compared to Ondansetron and Dexamethasone for Prophylaxis of Postoperative Vomiting in Children Undergoing Ambulatory Surgery: Clinical Trial Randomized, Double Blind, Placebo-controlled
Brief Title: Dexamethasone Compared to Ondansetron and Dexamethasone for Prophylaxis of Postoperative Vomiting in Children
Acronym: vomiting
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto Materno Infantil Prof. Fernando Figueira (Other)
Collaborators: Universidade Federal de Pernambuco (Other)
Responsible Party: Flavia Orange, Instituto Materno Infantil Prof. Fernando Figueira
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: 231/10
Record Dates: First submitted 2011-02-15; First posted 2011-02-16 (Estimated); Last update posted 2011-08-03 (Estimated); Status verified 2011-07

CONDITIONS: Vomiting Postoperative
Keywords: Nausea and Vomiting; Vomiting; Postoperative; Anesthesia
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Nausea; Vomiting | interventions — Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexamethasone (Placebo Comparator): Children randomized to this group received a 10 ml syringe containing dexamethasone (0.15 mg / kg) at the beginning of the procedure.
  Interventions: Drug: Dexamethasone
- Dexamethasone and ondasetron (Placebo Comparator): Children randomized to this group received a 10 ml syringe containing dexamethasone (0.15 mg / kg dose of 5mg ceiling) and ondansetron (0.1 mg / kg dose of 4mg ceiling)at the beginning of the procedure.
  Interventions: Drug: Dexamethasone and ondasetron

INTERVENTIONS:
Drug: Dexamethasone and ondasetron — Patients will receive ondansetron (0.1 mg / kg dose of 4mg cap) associated with dexamethasone (0.15 mg / kg dose of 5mg ceiling) or dexamethasone (0.15 mg / kg) or placebo
  Other Names: Decadron and nausedron
  Arms: Dexamethasone and ondasetron
Drug: Dexamethasone — Children were randomized to this group ni initiate proceedings with a 10ml syringe containing dexamethasone (0.15 mg / kg dose of 5mg ceiling)
  Other Names: Decadron
  Arms: Dexamethasone

SUMMARY:
The majority of pediatric surgery takes place in an outpatient basis. The occurrence of postoperative vomiting can lead to a delay in hospital discharge. However, the use of postoperative vomiting prophylaxis exposes patients unnecessarily to the drugs side effects and also raises the final costs of the surgical procedure. The Objective our study is Compare the incidence of postoperative vomiting between children who received dexamethasone, dexamethasone plus ondansetron or placebo for anti-emetic prophylaxis during outpatient surgery. This is a randomized, double blind, placebo-controlled study to comparing the use of dexamethasone, dexamethasone plus ondansetron and placebo for postoperative vomiting prophylaxis in children submitted to general anesthesia. Data analysis will be used is Fisher's exact test for the categorical variables and the Anova test for numerical variables as they presented Gaussian variation. The study used a significance level of 5%.

DETAILED DESCRIPTION:
The investigators know that a large number of pediatric surgeries are performed on an outpatient basis and the occurrence of nausea and vomiting after surgery can lead to delayed discharge and increased hospital costs. Based on this fact, the investigators find it relevant to determine the incidence of postoperative vomiting in pediatric surgery patients to assess the need for antiemetic prophylaxis in this study population being developed in the surgical ward of the Hospital das Clinicas - Federal University of Pernambuco (HC-UFPE ).

The study will be conducted from March 2011 to September 2011.Pacientes pediatric ASA I and II underwent surgery in the pediatric surgical ward of the HC-UFPE.

The sample size calculation was performed in the program StatCalc Epi-Info 6.04d, based on data from relevant literature and determined the presence of 44 patients in each of the three groups, totaling 132 patients in the study.

Patients will be recruited in the preparation room anesthetic in surgical clinics of the Hospital for three shifts of existing pediatric surgery. After evaluation of each patient and then filled the criteria of inclusion and exclusion, those responsible will be informed about the procedures being undertaken and the possible consequences of their participation in research.

Only after signing an informed consent by the person responsible will be held the allocation of patients into three groups, after opening the sealed envelope containing the selected group for that participant. These envelopes are previously prepared by a person outside the research.

Therefore, the researcher has no prior knowledge of the group selected for the participant at the time of the consent solicitation.

At the end of the study will fill a flowchart with the profile of the trial, including the total number of patients, the number of eligible patients, the number of those who were offered participation in the study, the number of denied and his reason the number of patients who agreed to participate. The latter will be known only after statistical analysis Randomization to each specific group will be held in accordance with a table of random numbers previously generated computer (Random Allocation Software 1.0, 2004).

Independent variable

* Use of dexamethasone and ondansetron, or dexamethasone or placebo only

Dependent Variables

* Incidence of postoperative vomiting;
* The need for antiemetic therapy in the recovery room post-anesthesia unit (PACU)
* Length of stay in PACU
* Delaying Hospital discharge All patients and their caregivers will be duly informed of the research objectives and will be included in the study only if they agree to participate and sign the Deed of Consent. The project was designed following the recommendations of Resolution 196/96 of the National Health Council and the Declaration of Helsinki for research involving human subjects (2000). In addition, the project was submitted to the Ethics Committee of the Hospital das Clinicas-UFPE and approved.

Patients will receive all information regarding the advantages and disadvantages of this technique, being safeguarded the right to refuse to participate. The researchers will undertake to publish the study, regardless of the outcome.

ELIGIBILITY:
Inclusion Criteria:

* ASA I or II
* Patients aged between 1 and 10 years old
* Patients undergoing general anesthesia for surgical repair of hernia, cryptorchidism and phimosis

Exclusion Criteria:

* Officials who refused to sign the consent form
* ASA ≥ III
* History of allergy to dexamethasone and/or ondansetron
* Patients taking opioids preoperatively
* Patients using antiemetic drugs preoperatively
* Patients with vomiting preoperatively

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 134 (Actual)
Dates: Start 2011-03; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Postoperative vomiting | The incidence of vomiting is seen in the anesthesia recovery room and 24 hours by phone
  Compare the incidence of vomiting in children who received dexamethasone or dexamethasone combined with ondansetron or placebo for antiemetic prophylaxis in ambulatory surgery.

SECONDARY OUTCOMES:
delayed discharge | In-room post-anesthesia recovery
  * Determine the relationship between the incidence of vomiting and the presence or absence of risk factors (duration ≥ 30 minutes of surgery, age ≥ 3 years and positive history in their own or relatives of postoperative vomiting).
  * To determine the association between pain in the immediate postoperative period and the incidence of postoperative vomiting
  * To determine the association between postoperative vomiting and delayed discharge

CONTACTS AND LOCATIONS:
Overall Officials: Flavia Orange, Investigator, Principal Investigator — Universidade Federal de Pernambuco